CLINICAL TRIAL: NCT02073799
Title: Change in Storage Symptoms Following Laser Prostatectomy: Comparison Between Potassium-titanyl-phosphate Photoselective Vaporization of the Prostate (PVP) and Holmium Laser Enucleation of the Prostate (HoLEP)
Brief Title: Storage Symptom After Laser Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LaserP1
Record Dates: First submitted 2014-02-23; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Photoselective vaporization of the prostate: Patients who underwent photoselective vaporization of the prostate for prostatic hyperplasia and in whom 12-months follow-up data were available
  Interventions: Procedure: Laser prostatectomy (Photoselective vaporization of the prostate or Holmium laser enucleation of the prostate)
- Holmium laser enucleation of the prostate: Patients who underwent holmium laser enucleation of the prostate for prostatic hyperplasia and in whom 12-months follow-up data were available
  Interventions: Procedure: Laser prostatectomy (Photoselective vaporization of the prostate or Holmium laser enucleation of the prostate)

INTERVENTIONS:
Procedure: Laser prostatectomy (Photoselective vaporization of the prostate or Holmium laser enucleation of the prostate)

SUMMARY:
Recent literature indicated that postoperative storage symptoms after Photoselective vaporization of the prostate (PVP) or holmium laser enucleation of the prostate (HoLEP) were often reported and generally more common than after transurethral prostatectomy (TURP). However, almost all literature focused on postoperative urgency or dysuria immediately after PVP or HoLEP. Thus, there has been a scarcity of data on serial changes of storage symptoms in the postoperative period after PVP or HoLEP and data on predicting factors that influence improvement in storage symptoms postoperatively. The aim of this study was to compare serial changes of postoperative storage symptoms between PVP and HoLEP, and to identify the predictors that influence improvement of storage symptoms postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of prostatic hyperplasia
* underwent photoselective vaporization of the prostate or holmium laser enucleation of the prostate
* 12-months follow-up data were available

Exclusion Criteria:

* previous diagnosis of urethral stricture, prostate carcinoma, and neurogenic bladder disease

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent photoselective vaporization of the prostate or holmium laser enucleation of the prostate and in whom 12-months follow-up data were available
Sampling Method: Non-Probability Sample
Enrollment: 486 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
the subtotal storage symptom score of the International Prostate Symptom Score (IPSS) | 12 months after surgery
  a reduction by ≥ 50% of the subtotal storage symptom score according to the International Prostate Symptom Score (IPSS) after the surgery compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Seoul National University Hospital, Seoul, Seoul, South Korea